CLINICAL TRIAL: NCT03129282
Title: A Feasibility Study on Integrating Home-based Metacognitive Therapy for Anxiety and Depression in the Cardiac Rehabilitation Pathway (PATHWAY STUDY WS3)
Brief Title: Pathway Study WS3 - Home Based Metacognitive Therapy for Cardiac Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Greater Manchester Mental Health NHS Foundation Trust (Other); University of Liverpool (Other)
Responsible Party: Principal Investigator, Adrian Wells, Professor, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 186990 (RP-PG-1211-20011)
Record Dates: First submitted 2017-04-11; First posted 2017-04-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Depression; Anxiety; Cardiac Rehabilitation; Psychological Distress
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants allocated to the "control" group will receive treatment as usual for cardiac rehabilitation
- Intervention (Active Comparator): Participants allocated to the "intervention" group will receive treatment as usual for cardiac rehabilitation plus the home-based metacognitive therapy (Home-MCT)
  Interventions: Other: Home-based Metacognitive Therapy (Home-MCT)

INTERVENTIONS:
Other: Home-based Metacognitive Therapy (Home-MCT) — Home-based metacognitive therapy (Home-MCT) is a facilitated self-help manual comprising six modules which participants will complete at their own pace over approximately 6 weeks. Participants will have an initial appointment with a Home-MCT trained cardiac rehabilitation staff members (face to face or by telephone). In addition, they will receive two telephone calls from trained cardiac rehabilitation staff members over the course of the intervention to offer support with completing the modules of the self-help manual.
  Arms: Intervention

SUMMARY:
Depression and anxiety are highly prevalent in people with heart disease, causing immense human and economic burden. Available pharmacological and psychological interventions have limited efficacy and the needs of these patients are not being met in cardiac rehabilitation services despite emphasis in key NHS policy.

Extensive evidence shows that a particular style of thinking dominated by rumination (dwelling on the past) and worry maintains emotional distress. A psychological intervention called metacognitive therapy (MCT) that reduces this style of thinking alleviates depression and anxiety in mental health settings.

This is a single-blind feasibility randomised controlled trial of metacognitive therapy delivered in a home-based format (Home-MCT). The aim of the study is to evaluate the acceptability and feasibility of integrating Home-MCT into cardiac rehabilitation services and to provide provisional evidence of effectiveness and cost-effectiveness on Home-MCT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are referred to the CR pathway who meet Department of Health (DoH) and/or British Association for Cardiovascular Prevention and Rehabilitation (BACPR) CR eligibility criteria:

   * Acute coronary syndrome used for any condition brought on by sudden, reduced blood flow to the heart
   * Following revascularisation is the restoration of perfusion to a body part or organ that has suffered ischemia
   * Stable heart failure
   * Stable angina is chest pain or discomfort that most often occurs with activity or stress
   * Following implantation of cardioverter defibrillators/cardiac resynchronisation devices
   * Heart valve repair/replacement
   * Heart transplantation and ventricular assist devices
   * Adult congenital heart disease identified in adulthood
   * Other (atypical heart presentation: nausea, dizziness, lower chest discomfort, upper abdominal pressure or discomfort that feels like indigestion and upper back pain)
2. A score of ≥ 8 on either the depression or anxiety subscale of the Hospital Anxiety and Depression Scale
3. Minimum of 18 years old
4. Competent level of English language skills

Exclusion Criteria:

1. Cognitive impairment which precludes informed consent or ability to participate
2. Acute suicidality
3. Active psychotic disorders (i.e., two [or more] of the following: delusions, hallucinations, disorganized speech, grossly disorganized or catatonic behaviour, negative symptoms).
4. Current drug/alcohol abuse (A maladaptive pattern of drinking, leading to clinically significant impairment or distress)
5. Concurrent psychological intervention for emotional distress that is not part of usual care
6. Antidepressant or anxiolytic medications initiated in the previous 8 weeks
7. Life expectancy of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Acceptability | From the completion of the manual till 4 months
  Acceptability of the intervention is defined as the completion of the first 4 modules of the Home-MCT manual, which includes 6 modules in total. Acceptability will be expressed as a % of all patients randomised to the treatment arm, minus deaths. This will be compared to the % of controls (minus deaths) who complete the 4-month follow up.

SECONDARY OUTCOMES:
Change in the Hospital Anxiety and Depression Scale (HADS) | Baseline, 4 months follow up, 12 months follow up
  The HADS is a 14-item self-report scale assessing anxiety and depression
Metacognitions Questionnaire 30 (MCQ-30) | Baseline, 4 months follow up, 12 months follow up
  The MCQ-30 is a 30-item self-report scale that measures: a) Lack of Cognitive Confidence, b) Positive Beliefs about Worry, c) Cognitive Self-Consciousness, d) Negative Beliefs about Uncontrollability and Danger, and e) Need to Control Thoughts
Cognitive Attentional Syndrome Scale (CAS-1) | Baseline, 4 months follow up, 12 months follow up
  The CAS-1 is a 10-item self-report measure assessing: a) the degree to which individuals have been dwelling on or worrying and/or focusing attention on threats, b) strategies used to cope with negative feelings and thoughts, and c) the degree to which individuals hold positive and negative metacognitive beliefs about worry
Impact of Events Scale - Revised (IES-R) | Baseline, 4 months follow up, 12 months follow up
  The IES-R is a 22-item self-report measure that assesses subjective distress caused by traumatic events
Health Related Quality of Life (EQ-5D) | Baseline, 4 months follow up, 12 months follow up
  The ED-5D is a standardised questionnaire for use as a measure of health status. It assesses: a) mobility, b) self-care, c) usual activities, d) pain/discomfort, and e) anxiety/depression, and the overall health status
Economic Patient Questionnaire (EPQ) | Baseline, 4 months follow up, 12 months follow up
  The EPQ assesses the services the patients have used as part of their health and social care
Credibility questionnaire (regarding the Home-MCT intervention) | From the completion of the introduction of the Home-MCT manual up to 2 weeks
  This is a 3-item self-report questionnaire assessing Home-MCT credibility to reduce psychological distress
Adherence questionnaire (regarding the Home-MCT intervention) | From the completion of the manual up to 4 months
  This is a 6-item self-report questionnaire assessing adherence to Home-MCT
Qualitative interviews with intervention patients to identify enablers and barriers to recruitment and engagement with the intervention (Home-MCT) | Up to 2 weeks before receiving the intervention and up to 1 month after the completion of the intervention
  Interviews are aimed to explore patient's experiences of going through the Home-MCT intervention

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Wells, PhD, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Bolton NHS Foundation Trust, Bolton
  - Aintree Liverpool NHS Foundation Trust, Liverpool

REFERENCES:
- [Result] Wells A, Reeves D, Heal C, Fisher P, Doherty P, Davies L, Heagerty A, Capobianco L. Metacognitive therapy self-help for anxiety-depression: Single-blind randomized feasibility trial in cardiovascular disease. Health Psychol. 2022 May;41(5):366-377. doi: 10.1037/hea0001168. PMID 35467904
- [Derived] Wells A, Reeves D, Heal C, Davies LM, Shields GE, Heagerty A, Fisher P, Doherty P, Capobianco L. Evaluating Metacognitive Therapy to Improve Treatment of Anxiety and Depression in Cardiovascular Disease: The NIHR Funded PATHWAY Research Programme. Front Psychiatry. 2022 Jun 3;13:886407. doi: 10.3389/fpsyt.2022.886407. eCollection 2022. PMID 35722590
- [Derived] Wells A, McNicol K, Reeves D, Salmon P, Davies L, Heagerty A, Doherty P, McPhillips R, Anderson R, Faija C, Capobianco L, Morley H, Gaffney H, Heal C, Shields G, Fisher P. Metacognitive therapy home-based self-help for cardiac rehabilitation patients experiencing anxiety and depressive symptoms: study protocol for a feasibility randomised controlled trial (PATHWAY Home-MCT). Trials. 2018 Aug 16;19(1):444. doi: 10.1186/s13063-018-2826-x. PMID 30115112
- See also: Web-site with details about the study — http://www.adept-ru.com